CLINICAL TRIAL: NCT06774703
Title: Nemaline Myopathy Clinical Research Network (NM-CTRN)
Status: Not yet recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: A Foundation Building Strength (Other)
Responsible Party: Principal Investigator, Carolina Tesi-Rocha, Clinical Professor, Stanford University
Other Study IDs: 72180
Record Dates: First submitted 2024-03-14; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Nemaline Myopathy
Keywords: Neuromuscular disease; Observational study; Congenital myopathy; Nemaline rod
MeSH Terms: conditions — Myopathies, Nemaline; Neuromuscular Diseases; Myotonia Congenita

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Plasma, serum and DNA samples will be retained. Exact amounts will depend on age of participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Individuals with Nemaline Myopathy: All participants in the study will have a diagnosis of Nemaline Myopathy, with either a pathogenic or likely pathogenic mutation in ACTA1 (AD) or NEB (AR). Participants can be either ambulatory or non-ambulatory and must be between the ages of 0-18.

SUMMARY:
The goal of this study is to establish a research network to help define the natural disease history and clinical outcome measures for Nemaline Myopathy (NM).

DETAILED DESCRIPTION:
The long-term aim of this study is to incorporate these outcome measures into clinical trials for NM therapies. Outcome measures to be assessed will be dependent on the participant's age and functional status. Follow-up visits will be conducted either every 3 or 6 months, dependent on age, for a total of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* 0-18 years of age at recruitment
* Confirmation of Nemaline Myopathy (pathogenic or likely pathogenic mutations in ACTA1 (AD) or NEB (AR)
* Patient and/or parent or legal guardian must be willing and able to provide informed consent

Exclusion Criteria:

* Clinically significant medical finding on the physical examination, other than NM, that the Investigator deems unsuitable for participation in and/or completion of the study procedures
* Any confirmed chronic or acute condition or disease affecting any system(s), which could interfere with the results of the study and/or the compliance with the study procedures. This will be subject to the clinical judgement of the Principal Investigator (PI)
* Participants of ongoing (interventional) clinical trials that assess the efficacy of potential treatments will be excluded
* Safety concerns

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be identified through several sources. The primary source will be through our NM-CRN MDA care center network. Participants will also be recruited through the CMDIR and the Beggs Laboratory. Information regarding the study will be disseminated to all MDA clinics through the MDA website and via email to clinic directors. In addition, the study will advertised to families through A Foundation Building Strength, which maintains a patient information website and newsletter.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Validate the change over 36 months using the Alberta Infant Motor Scale (AIMS) Score | 36 months
  The AIMS is a standardized tool used to assess a child's gross motor development in four positions: prone, supine, sitting, and standing. Percentile scores are given from 0-100, with higher percentiles representing higher motor function.
Validate the change over 36 months using the Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP-INTEND) | 36 months
  The CHOP-INTEND assesses a child's ability to move their body in a lying down position, supported sitting, and assisted rolling through 16 items.
Validate the change over 36 months using the Hammersmith Infant Neurological Examination Section 2 (HINE-2) | 36 months
  This is a 37-item measure of infant developmental motor milestones divided into the following categories: neurological examination, developmental milestones and behavioral scale, and state of consciousness. Scores for individual categories will be combined into a composite score.This will be performed in participants aged 0-24months. Scores are interpreted in relation to optimality scores and cut-off scores for the participant's age. Higher scores represented higher function.
Validate the change in 32-item Motor Function Measure (MFM32) Scale Score | 36 months
  This motor function assessment consists of 32 items organized in three dimensions: standing position and transfers, axial and limb proximal motor function, and limb distal motor function. Total scores are given between 0-100, with 0 indicating severe functional impairment and 100 indicating no functional impairment.
Change in Peabody Developmental Motor Scales (PDMS-3) Scale Score | 36 months
  This is used to measure various motor abilities in young children. Four types of normative scores are yielded: age equivalents, percentile ranks, subtest scaled scores, and composite index scores. Age equivalents are indexes of relative standing that translate subtest raw scores into motor ages. Percentiles provide the examiner with an index that is easily understood. Subtest scaled scores are based on a distribution having a mean of 10 and a standard deviation of 3. Composite indexes are based on a distribution with a mean of 100 and a standard deviation of 15. Higher scores indicate higher level of function.
Change in ambulation over 36 months as measured by the 10 meter walk (m/s). | 36 months
  This test measures the time taken for a participant to walk 10 metres as quickly and safely as possible. This will be performed in ambulatory participants aged 2 years and older.
Change in ambulation over 36 months as measured by the 6 Minute Walk Test | 36 months
  This is a measure of how far a participant can walk along a track in 6 minutes. This will be performed in ambulatory participants aged 5 years and older.
Change in respiratory function over 36 months as measured by spirometry, specifically the supine forced vital capacity (FVC). | 36 months
  This is a measure (% predicted) of the maximum amount of air that can be forcibly exhaled from your lungs after taking the deepest breath possible. This will be performed in participants aged 5 years and older.

SECONDARY OUTCOMES:
Change in muscle thickness of lower extremity muscles over 36 months as measured by muscle ultrasound. | Baseline through month 36
  This will be conducted in a subset of participants aged >5 years.
Skin Biopsy (optional) | Baseline through month 36
  This optional outcome measure involves a one-time removal of three to four 2mm pieces of skin from one body site.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Tesi-Rocha, MD, Principal Investigator — Stanford University; Tina Duong, PT, PhD, Principal Investigator — Stanford University; John W Day, MD, PhD, Principal Investigator — Stanford University; Leslie Hayes, MD, Principal Investigator — Boston Children's Hospital; Alan Beggs, PhD, Principal Investigator — Boston Children's Hospital; Jim Dowling, MD, PhD, Principal Investigator — The Hospital for Sick Children; Richard Finkel, MD, Principal Investigator — St Jude Children's Hospital; Carsten Bonnemann, MD, PhD, Principal Investigator — National Institutes of Health (NIH); Kaitlin Batley, MD, Principal Investigator — UT Southwestern Medical Centre
Locations (6):
- United States (5):
  - Stanford University/Lucile Packard Children's Hospital, Palo Alto, California
  - National Institute of Health, Bethesda, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - UT Southwestern Medical Centre/Children's Health Dallas, Dallas, Texas
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes